CLINICAL TRIAL: NCT06689891
Title: Utilizing Remote, Video-Based Pelvic Floor Muscle Therapy: A Feasibility Trial
Brief Title: Video-Based Pelvic Floor Muscle Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2000037163
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pelvic Floor Disorder; Pelvic Floor Muscle Exercise
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Intervention Model Description: Study population will include patients who have an indication for referral for pelvic floor rehabilitation (PFR).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Video-based pelvic floor muscle therapy (PFMT) (Experimental): Patients will complete a series of surveys before and after the intervention. They will complete 8 weeks of video-based PFMT with an initial and final in-person session with a pelvic floor therapist.
  Interventions: Device: Pelvic Floor Muscle Therapy Website

INTERVENTIONS:
Device: Pelvic Floor Muscle Therapy Website — 8-week video-based, self-directed PFMT course

SUMMARY:
This study is a feasibility, pilot trial of remote, video-based pelvic floor muscle therapy (PFMT) for patients with pelvic floor disorders, including pelvic organ prolapse, urinary incontinence and anorectal dysfunction. PFMT has been shown to improve these symptoms in multiple studies.

DETAILED DESCRIPTION:
This will be a feasibility and acceptability trial of a novel remote, web-accessible PFMT curriculum, designed by pelvic floor physical therapists.

Patients will be expected to complete a 5-10-minute survey at initial enrollment. They will have one in-person session with a pelvic floor therapist prior to starting the 8-week video-based PFMT course. Afterwards, they will have a final in person session with a pelvic floor therapist along with a final set of surveys that should take an estimated 10-15 minutes.

The primary objective is to the determine the feasibility and accessibility of using a video-based PFMT for patients with pelvic floor dysfunction.

The secondary objective is to determine whether video-based PFMT can improve symptomatology and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pelvic floor dysfunction with referral for PFR
* English-speaking

Exclusion Criteria:

* Unable to access web-based videos
* Unable to speak English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale (SUS) Score | 8 weeks
  The SUS is a 10-question survey that measures how easy a product or system is to use. Total score range from 0-100 with higher scores indicating better usability.
Percentage of participants video completion | 8 weeks
  Percentage of participants that complete at least 80% of the videos
Change in graded evaluation of exercises by pelvic floor therapist | baseline and 8 weeks
  Participants will be assessed and graded and by the pelvic floor physical therapist as below: 1 - cannot perform exercise, 2 - can partially perform exercise (needs some cueing and assistance), 3 - can independently perform exercise
Adverse Events | up to 8 weeks
  Number of participants that experience at least one adverse event.

SECONDARY OUTCOMES:
Short Form-12 (SF-12) | baseline and week 9
  The SF-12 is an abbreviated version of the SF-36. The SF-12 is a validated survey that assesses a patient's health related quality of life across eight domains. The total score range is 0-100 with a physical component summary and a mental component summary. A higher score indicates better health for each of those components.
Cleveland Clinic Incontinence Score (CCIS) | baseline and week 9
  The CCIS is a health-related quality of life measure that assesses how often and to what degree incontinence affects a person's life. The total score ranges from 0 to 20, with higher scores indicating higher levels of incontinence.
Patient Assessment of Constipation Symptoms (PAC-SYM) | baseline and week 9
  The PAC-SYM is a questionnaire used to assess the severity of constipation symptoms in adults. Total score range 0-4 with higher scores indicating more severe constipation.
International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) | baseline and week 9
  The ICIQ-SF is a brief patient-completed questionnaire that measures the impact of urinary incontinence (UI) on quality of life (QoL). The ICIQ-UI SF is scored on a scale of 0-21. A score of zero means no urine leakage and no impact on QoL.
Pelvic Organ Prolapse Symptom Score (POP-SS) | baseline and week 9
  The POP-SS is a questionnaire that measures the severity of pelvic organ prolapse symptoms. The total score ranges from 0-28, with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No